CLINICAL TRIAL: NCT06848257
Title: The Effect of Postural Exercises on the Perception of Verticality in Parkinson's Disease
Brief Title: Posture Exercises in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Aysegul Gokturk Usta, Asistant Professor, Yuksek Ihtisas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/03/10
Record Dates: First submitted 2025-01-14; First posted 2025-02-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Parkinson
Keywords: Parkinson; Postural exercises; Verticality; Position sense
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinic research (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — postural exercises

SUMMARY:
The research was planned as a quasi-experimental study to investigate the effects of postural exercises on body image and neck and trunk position sense in Parkinson's patients.

It was decided to conduct the study with Parkinson's patients over the age of 50 who applied to the neurology clinic. After the power analysis for the research, it was planned to reach 36 participants. Participants' consent to participate in the study will be obtained through the Informed Volunteer Consent Form prepared by the researchers. Demographic information of participants who consent to participate in the study will be collected. Then, the disease levels and severity of the participants will be determined using the Modified Hoehn Yahr Staging Scale and the Unified Parkinson's Disease Assessment Scale. Subjective Visual Vertical Perception, Subjective Postural Perception and Subjective Haptic Perception evaluations to evaluate the body image of patients; Clinometer application and neck and trunk proprioception evaluations will be applied as preliminary tests to evaluate neck and trunk position sense. Posture exercises planned by the researchers will be applied to the participants, whose pre-tests are completed, three days a week for eight weeks. Preliminary tests performed after eight weeks of exercise will be repeated. All data obtained will be recorded in the Participant Data Record form. Differences in changes in tests performed at eight-week intervals will be investigated with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Being over 50 years old,
* Being diagnosed with Parkinson's disease by a physician,
* Stage 1-4 according to the modified Hoehn-Yahr staging scale
* Having received 24≥ from the Mini Mental test

Exclusion Criteria:

* Presence of another accompanying neurological disease,
* Having significant musculoskeletal system problems,
* Having any known cognitive problem or having a score of ≤23 on the Mini Mental Test

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics of the individuals participating in the study | All evaluations will be done before and after the treatment (8 weeks)
  Demographic information of the patients such as age(years), height (in meters) and weight (in kilograms) and education level (primary school, secondary school, high scool, etc) will be recorded. Weight and height will be used to calculate Body mass index (BMI) (kg/m^2). BMI will be used to compare body compositions of patients. Mini Mental Test; used to evaluate cognitive performance.Those who score 24 points or above on the test (being able to understand and apply the given commands) will be included in the study.
Evaluations about Parkinson's disease | All evaluations will be done before and after the treatment (8 weeks)
  Disease staging of individuals will be done with the Modified Hoehn and Yahr Scale (MH&YS). In this scale, patients are divided into 5 main categories according to their level of independence status.According to the scale, patients who can walk without support (at most stage 3) will be included in the study. And disease severity will be measured by Unified Parkinson's Disease Rating Scale(UPDRS) .The scale consists of 4 sections to evaluate different systems. These are; emotion-thought (total 16 points), motor (total 92 points), daily life (total 52 points), treatment and complications (total 23 points). Each evaluation step is scored between 0 and 4. A low total score indicates that the severity of the disease is low, while an increase in the total score indicates that the disease is severe.
Subjective verticality perception evaluations | All evaluations will be done before and after the treatment (8 weeks)
  Assessment of Subjective Vertical Perception:The Bucket Test evaluates subjective visual verticality by having participants align a vertical line inside a bucket without external visual cues.For Postural Vertical, an inclinometer measures deviations as participants adjust their torso to perceived verticality in 0°, 30° right, and 30° left positions.Haptic Vertical is tested by blindfolded participants aligning a rod to reference angles (0°, 45° left, 45° right).Scored by taking the absolute value of the deviations from three trials
proprioception evaluations | All evaluations will be done before and after the treatment (8 weeks)
  Position Sense (proprioception) is assessed by repositioning the neck (C7) and trunk (L1) to a 30° flexion target. Scored by taking the absolute value of the deviations from three trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no reason.